CLINICAL TRIAL: NCT01403493
Title: A Comparison of a Short Nurse Based and a Long Multidisciplinary Version of Structured Patient Education in Irritable Bowel Syndrome.
Brief Title: Multidisciplinary Versus a Nurse Based Patient Education For Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Magnus Simren, Sahlgrenska University Hospital, Gothenburg, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-487-02 amendment
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Patient education
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary patient education (Active Comparator): A multidisciplinary (nurse, gastroenterologist, dietician, physiotherapist, psychologist) group education with six sessions for patients with IBS.
  Interventions: Behavioral: Patient education
- Nurse based patient education (Active Comparator): A nurse based patient education with three sessions for patients with IBS.
  Interventions: Behavioral: Patient education

INTERVENTIONS:
Behavioral: Patient education

SUMMARY:
In this randomized controlled study in patients with irritable bowel syndrome (IBS), the investigators plan to compare the effects of a multidisciplinary structured patient group education with a compressed nurse based structured patient group education. The effects of the interventions on gastrointestinal (GI) and psychological symptom severity, knowledge and quality of life will be assessed with validated questionnaires at baseline and 3, 6 and 12 months after the intervention.

DETAILED DESCRIPTION:
In this randomized controlled study in patients with irritable bowel syndrome (IBS) we plan to compare the effects of a multidisciplinary, structured patient group education with a compressed, nurse based, structured patient group education. We plan to include men and women 18 to 70 years old, with IBS according to the Rome II criteria, who are referred from physicians in primary care and secondary/tertiary care to participate in the study. The education will be held at the GI out patient clinic at Sahlgrenska University hospital in Gothenburg. The patients will be informed about the positive results obtained in previous studies with different educational interventions. Patients with an organic GI disease and/or with another disease potentially affecting the GI symptoms are excluded. Likewise, patients with a severe psychiatric disease are excluded due to potential problems to participate in a group intervention. In order to allocate an equal number of patients to both of the interventions during the study, a number of up to 20 patients will be included in a block. The patients will be randomly divided into two groups with an equal number of patients in each group. The groups will then be randomized 1:1 to either start the multidisciplinary or the nurse based education within two to three weeks. The effects of the interventions on GI and psychological symptom severity, knowledge and quality of life will be assessed with validated questionnaires at baseline and 3, 6 and 12 months after the intervention:

1. Perceived knowledge about IBS
2. IBS Severity Scoring System (IBS-SSS)
3. IBS Quality of Life (IBSQOL)
4. Visceral Sensitivity Index (VSI)

4. The Hospital Anxiety and Depression Scale (HAD)

The interventions:

The education is designed based on the self-efficacy theory , and the general theory of nursing. Moreover, the education is performed based on a biopsychosocial model considered to be important in functional GI disorders. The multidisciplinary education consists of six sessions held once per week in a group setting with eight to ten patients in each group. Five different health care professionals (nurse, gastroenterologist, dietician, physiotherapist and psychologist) are involved in the education, in order to cover a wide spectra of issues related to IBS. Each of the professionals will hold one session for two hours where a lot of space is given for discussion in the group. This intervention has been described in detail previously (Ringström et. al. BMC Gastroenterol 2009;9:10).

The nurse based education consists of three sessions held ones per week in a group setting with eight to ten patients in each group. A nurse, special trained in gastroenterology, is involved in this education, which covers the same spectra of issues related ti IBS as the multidisciplinary version.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 70 years old, with IBS according to the Rome II criteria.
* Written informed consent

Exclusion Criteria:

* An organic GI disease and/or with another disease potentially affecting the GI symptoms.
* Severe psychiatric disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effect on GI symptoms as measured by IBS-SSS and satisfactory relief of IBS symptoms | Change from Baseline in GI Symptom severity and satisfactory relief of IBS symptoms at 3, 6 and 12 months.

SECONDARY OUTCOMES:
Effects on Quality of life (IBSQOL), Psychological symptoms (HAD), GI specific anxiety (VSI) and knowledge about IBS | Change from Baseline in quality of life, psychological symptoms and knowledge at 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simren, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden